CLINICAL TRIAL: NCT04408144
Title: Effectiveness of Treatment With Additional Dydrogesterone (Duphaston) to the Standard Luteal Phase Support After Fresh Embryo Transfer: a Prospective Randomized Controlled Trial.
Brief Title: Addition of Dydrogesterone to the Luteal Phase Support After Fresh Embryo Transfer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laniado Hospital (Other)
Responsible Party: Principal Investigator, Amir Weintraub, Director, IVF Unit, Laniado Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0003-20-LND
Record Dates: First submitted 2020-05-12; First posted 2020-05-29 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Infertility; IVF
MeSH Terms: conditions — Infertility | interventions — Dydrogesterone; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- StudyGroup (Experimental): Patients will receive an addition of dydrogesterone (Duphaston) to the standard treatment for luteal phase support
  Interventions: Drug: Dydrogesterone 10mg Oral Tablet
- Control Group (No Intervention): Patients will receive the standard treatment for luteal phase support without Dydrogesterone

INTERVENTIONS:
Drug: Dydrogesterone 10mg Oral Tablet — oral 10mg dydrogesterone (Duphaston) 2 times daily
  Arms: StudyGroup

SUMMARY:
Randomized controlled study, open label to compare effectiveness of addition of dydrogesterone 20mg to the standard luteal phase support treatment after fresh embryos transfer.

DETAILED DESCRIPTION:
In the context of IVF treatment, it's a standard of care to use progesterone for endometrial synchronization and for luteal phase support after embryos transfer and until week 9-12 of pregnancy.

In Israel, as in most european countries, vaginal insert of Micronised Vaginal Progesterone (MVP) is mostly prescribed.

Dydrogesterone is a potent active progesterone receptor agonist that is well tolerated, orally administered and is considered to be sufficiently safe during pregnancy.

Based on recent publications, single oral dydrogesterone treatment seems to be a good option in clinical practice for luteal phase support in IVF cycles with fresh embryos transfer.

But, until now, there is no publication evaluating the effectiveness of an addition of Dydrogesterone to the standard of care.

The aim of the study is to compare effectiveness of addition of dydrogesterone 20mg to the standard luteal phase support treatment after fresh embryos transfer.

The trial is a randomized controlled study, open label. Participants will receive either standard treatment with an addition of oral 10mg dydrogesterone (Duphaston) 2 times daily or the standard treatment without Dydrogesterone, starting on the day of fresh embryos transfer until 10 weeks of gestation or until pregnancy test is negative.

Study participation will be proposed to every woman going through fresh embryos transfer in Laniado IVF unit, who meets the inclusion/exclusion criteria.

The investigators aim to include 150 patients in each arm of the study, during 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a documented history of infertility who underwent IVF with or without ICSI, going through embryos transfer (having in the past up to 2 previous embryos transfer) and who gave written informed consent.
* Body mass index ≥18 to ≤35 kg/m2
* LH, prolactin (PRL), testosterone and thyroid-stimulating hormone (TSH) within normal clinical limits or not considered clinically significant within 1 year prior to or at screening
* Normal transvaginal ultrasound at screening (or within 14 days prior to screening)
* Planning a transfer of 1 or 2 fresh embryos.

Exclusion Criteria:

* Previous participation in this trial
* Subjects with >2 unsuccessful IVF attempts
* Evidence of head, ear, eye, nose, throat, cardiovascular, respiratory, urogenital, gastrointestinal/hepatic, hematologic/immunologic, dermatologic/connective tissue, musculoskeletal, metabolic/nutritional, endocrine or neurologic/psychiatric disorders;
* Recent major surgery (within 3 months);
* Current or recent substance abuse, including that of alcohol and tobacco;
* History of chemotherapy;
* History of recurrent pregnancy loss (≥3 previous miscarriages)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 9 month
  The percentage of live newborns in the total cycles of treatment

SECONDARY OUTCOMES:
Presence of fetal heartbeats at 12 weeks of gestation | 12 weeks
  The percentage of pregnancies with heartbeats observed by ultrasound at 12 weeks in the total cycles of treatment
Frequency of positive pregnancy tests on Day 14 after embryo transfer | 14 days
Rates of obstetrical complications | 9 months
  Obstetrical complications during pregnancy and labor. Examples- abruptio placenta, First trimester bleeding, Preterm Prelabor Rupture Of Membranes (PPROM), preterm labor
Newborn outcomes | 1 year
  Appearance, Pulse, Grimace, Activity and Respiration (APGAR) score- between 0-10. 10 is the best outcome. 0 is the worst outcome.
Newborn Weight | 9 months
  in grammes
Rates of Newborn malformations | 1 year
  Abnormal findings of physical examination of the newborn

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 3 years
  Adverse Events (AES) and Serious Adverse Events (SAES) will be recorded during all the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Laniado Hospital, Netanya, Israel